CLINICAL TRIAL: NCT06408194
Title: Phase I/Ib Clinical Trial of Autologous CD22 Chimeric Antigen Receptor (CAR) T Cells Following Commercial CD19 CAR T Cells in Children and Young Adults With Recurrent or Refractory B Cell Malignancies
Brief Title: Autologous CD22 CAR T Cells Following Commercial CD19 CAR T Cells in B Cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-74214; NCI-2024-04331 (Other: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2024-04-22; First posted 2024-05-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Leukemia; Acute Lymphoblastic Leukemia
Keywords: KYMRIAH; CAR T; Tisagenlecleucel; Lymphodepletion
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lymphodepletion (Experimental): All enrolled participants will receive lymphodepletion followed by standard of care tisagenlecleucel infusion.
  Interventions: Drug: CD22CART infusion; Drug: Tisagenlecleucel

INTERVENTIONS:
Drug: CD22CART infusion — CD22CART will be administered after Standard of Care (SOC) administration of tisagenlecleucel.
Drug: Tisagenlecleucel — All enrolled participants will receive lymphodepletion followed by standard of care tisagenlecleucel infusion.
  Other Names: KYMRIAH

SUMMARY:
The primary purpose of this study is to determine safety, feasibility, and the Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D) of CD22 Chimeric Antigen Receptor T-Cell Therapy (CART) cells when administered 28 to 42 days after an infusion of a commercial CAR called Tisagenlecleucel, to children and young adults with relapsed or refractory B-cell leukemia.

DETAILED DESCRIPTION:
Primary Objectives:

Phase 1 portion (Safety lead-in):

Determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) dose of CD22CART in children and young adults with R/R CD19 and CD22 expressing B-cell malignancies administered after infusion of tisagenlecleucel according to FDA approved dose range.

Phase 1b portion (Expansion cohort) Establish the feasibility of delivering CD22CART following infusion of commercial tisagenlecleucel, administered per FDA approved Package Insert, in children and young adults with B cell malignancies.

Determine the safety of administering the RP2D of CD22CART 28 to 42 days after infusion of FDA approved commercial tisagenlecleucel in children and young adults with B cell malignancies.

Secondary Objectives:

1. Describe the clinical activity of serial infusion of tisagenlecleucel followed by CD22CART in children and young adults with R/R B-cell malignancies.
2. Assess the rate of ongoing B cell aplasia at 6 months after initial tisagenlecleucel infusion, when tisagenlecleucel is followed by serial CD22CART infusion within 42 days.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of histologically confirmed relapsed/refractory (R/R) B cell acute lymphoblastic leukemia (ALL)
2. Must be eligible to receive commercial KYMRIAH® (tisagenlecleucel) according to FDA approved package insert (refractory disease or in second or later relapse)
3. CD19 and CD22 expression must be demonstrated on malignant cells by immunohistochemistry or flow cytometry. CD19 and CD22 expression at any level of expression will be acceptable, as that is the standard for commercial KYMRIAH® (tisagenlecleucel) and the optimal level of CD22 expression is not well defined.
4. Age: ≥ 1 year of age and ≤ 25 years and 364 days of age at time of enrollment.
5. Performance Status: Participants > 16 years of age: Karnofsky ≥ 50%; Participants ≤ 16 years of age: Lansky scale ≥ 50%.
6. Normal Organ and Marrow Function

   * Absolute Neutrophil Count (ANC) ≥ 750/uL*
   * Platelet count ≥ 50,000/uL*
   * Absolute Lymphocyte Count ALC > 150/uL*
   * Adequate renal, hepatic, pulmonary and cardiac function defined as:

     * Baseline oxygen saturation > 92% on room air
     * Creatinine within ULN for age or Creatinine clearance (as estimated by Cockcroft Gault Equation) ≥ 60 mL/min
     * Total bilirubin ≤ 1.5 mg/dl, except in Participants with Gilbert's syndrome. [Elevations related to leukemia involvement of the liver will not disqualify a subject]
     * Alanine Transaminase (ALT) or Aspartate Aminotransferase (AST) ≤ 10 x ULN (except in Participants with liver involvement by leukemia)
     * Cardiac ejection fraction ≥ 40%, no evidence of pericardial effusion as determined by an Echocardiogram.
     * if these cytopenias are not judged by the investigator to be due to underlying disease (i.e. potentially reversible with anti-neoplastic therapy); A subject will not be excluded because of pancytopenia ≥ Grade 3 if it is due to disease, based on the results of bone marrow studies.
7. Participants with Central Nervous System (CNS) involvement or a history of CNS involvement are eligible only in the absence of neurologic symptoms that may mask or interfere with neurological assessment of toxicity
8. Participants who have undergone autologous SCT with disease progression or relapse following SCT are eligible. Participants with history of allogeneic SCT must be at least 100 days from SCT, have no evidence of Graft versus Host Disease (GvHD), and no longer taking immunosuppressive agents for at least 30 days prior to enrollment.
9. Females of child bearing potential and males of child fathering potential must be willing to practice birth control during and for 4 months post chemotherapy or for as long as Chimeric Antigen Receptor (CAR) T cells are detectable in peripheral blood.
10. Females of child bearing potential must have negative pregnancy test.
11. Must meet wash out period since prior therapies according to commercial KYMRIAH® (tisagenlecleucel) SOPs.
12. Must have recovered from acute side effects from prior therapy to meet eligibility.
13. If had prior CAR therapy, will be eligible if at least 30 days has elapsed prior to apheresis.
14. Ability to give informed consent. All Participants ≥ 18 years of age must be able to give informed consent. For participants <18 years old their legal authorized representative (LAR) (i.e. parent or guardian) must give informed consent. Pediatric participants will be included in age appropriate discussion and assent per institutional SOPs will be obtained for those > 7 years of age, when appropriate. If a minor becomes of age during participation of this study, he/she will be asked to reconsent as an adult.

    * A subject will not be excluded because of pancytopenia ≥ Grade 3 if it is felt by the investigator to be due to underlying disease.

Exclusion Criteria:

1. May not have Human Immunodeficiency Virus (HIV)/Hepatitis B (HBV) or Hepatitis C (HCV infection) or uncontrolled, symptomatic, intercurrent illness.
2. May not have hyperleukocytosis (≥ 50,000 blasts/μL) or rapidly progressive disease that in the estimation of the investigator and sponsor would compromise ability to complete study therapy.
3. May not have severe, immediate hypersensitivity reaction attributed to compounds of similar chemical or biologic composition to any agents used in study.
4. May not have active CNS disorder, or history of MI, cardiac angioplasty or stenting, unstable angina or other clinically significant cardiac disease with 12 months of enrollment.
5. May not have primary immunodeficiency or history of autoimmune disease (e.g. Crohns, rheumatoid arthritis, systemic lupus) requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The number of patients who experience dose limiting toxicities (Phase 1) | 28 days after single infusion of CD22 CAR T cells
  The number of patients who experience dose limiting toxicities within 28 days of administration of CD22 CART when given within 28-42 days of infusion of tisagenlecleucel
The number of patients who successfully receive infusion of CD22CART (Phase 1b) | within 42 days of infusion of tisagenlecleucel
  The number of patients who successfully receive infusion of CD22CART within 42 days of infusion of tisagenlecleucel

SECONDARY OUTCOMES:
Number of patients who have no evidence of leukemia | 28 days after single infusion of CD22 CAR T cells
  Number of patients who have no evidence of leukemia (complete response or complete response with incomplete count recovery) at Day 28 following CD22 CART infusion.
The number of patients who have B cell aplasia | 6 months following single infusion of CD22 CAR T cells and tisagenlecleucel
  The number of patients who have B cell aplasia 6 months following tisagenlecleucel and CD22 CART infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States